CLINICAL TRIAL: NCT03007342
Title: Effect of Amoxicillin/Clavulanic Acid Combination on Postoperative Endodontic Pain in Patients With Symptomatic Apical Periodontitis: A Randomized Controlled Trial
Brief Title: Effect of Amoxicillin/Clavulanic Acid Combination on Postoperative Endodontic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Gomaa, Post-graduate candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEBC-CU-2016-11-168
Record Dates: First submitted 2016-12-19; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Symptomatic Periapical Periodontitis
Keywords: Amoxicillin; clavulanic acid; Periapical periodontitis; Post-operative pain
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative | interventions — Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Oral tablet 1000 mg of Amoxicillin/ clavulanic acid combination every 12 hours for five days.
  Interventions: Drug: Amoxicillin/Clavulanate Potassium 875 mg-125 mg oral tablet
- control group (Placebo Comparator): Oral tablet placebo every 12 hours for five days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin/Clavulanate Potassium 875 mg-125 mg oral tablet
  Arms: Experimental group
Drug: Placebo
  Arms: control group

SUMMARY:
The aim of this prospective, randomized, placebo controlled study is to evaluate the effect of amoxicillin/clavulanic acid combination on post-operative pain and swelling in adult patient with symptomatic apical periodontitis.

DETAILED DESCRIPTION:
Medical and dental history will be obtained from all patients participating in this trial. Clinical and radiographic evaluation for each tooth included in this study will be recorded.

Clinical diagnosis of symptomatic apical periodontitis is to be confirmed.

After single-visit root canal treatment, eligible participants will be randomly assigned to one of the following groups: experimental group (taking oral tablet 1000 mg of Amoxicillin/ clavulanic acid combination) or control group (taking placebo tablet).

Each patient will receive a 7-day diary to record postoperative pain and swelling.In case of pain, the participant will be instructed to take an analgesic. Post-operative pain will be measured as a primary outcome on 11-point scale (NRS) at the following time points: 6, 12, 24, 48, 72 hours and 7 days. The occurrence of swelling will be reported by participant as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic apical periodontitis who do not have evidence of spreading infection or systemic involvement.
2. Mandibular posterior teeth with positive response to percussion.
3. Patients with non-contributory systemic condition.
4. Patients who can understand pain scales and able to sign informed consent.

Exclusion Criteria:

1. Patients allergic to penicillin.
2. Patients who have a draining sinus tract.
3. Retreatment cases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain. | Up to 7 days after endodontic treatment
  Post-operative pain will be measured by a numerical rating scale (NRS).

SECONDARY OUTCOMES:
Swelling | 7 days
  The occurrence of Swelling will be measured by a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gomaa, Postgraduate, Principal Investigator — Cairo University; khaled Ezzat, Professor, Study Chair — Cairo University; Suzan AW Amin, PhD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henry M, Reader A, Beck M. Effect of penicillin on postoperative endodontic pain and swelling in symptomatic necrotic teeth. J Endod. 2001 Feb;27(2):117-23. doi: 10.1097/00004770-200102000-00016. PMID 11491635
- [Background] Fouad AF, Rivera EM, Walton RE. Penicillin as a supplement in resolving the localized acute apical abscess. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1996 May;81(5):590-5. doi: 10.1016/s1079-2104(96)80054-0. PMID 8734709
- [Background] Cope A, Francis N, Wood F, Mann MK, Chestnutt IG. Systemic antibiotics for symptomatic apical periodontitis and acute apical abscess in adults. Cochrane Database Syst Rev. 2014 Jun 26;(6):CD010136. doi: 10.1002/14651858.CD010136.pub2. PMID 24967571
- [Background] Arteagoitia MI, Barbier L, Santamaria J, Santamaria G, Ramos E. Efficacy of amoxicillin and amoxicillin/clavulanic acid in the prevention of infection and dry socket after third molar extraction. A systematic review and meta-analysis. Med Oral Patol Oral Cir Bucal. 2016 Jul 1;21(4):e494-504. doi: 10.4317/medoral.21139. PMID 26946211